CLINICAL TRIAL: NCT02013830
Title: A Single-arm, Open-label Study of Avastin Plus Xeloda on Objective Treatment Response in Patients With Advanced or Metastatic Liver Cancer Who Have Had no Previous Cytotoxic Chemotherapy
Brief Title: A Study of Avastin (Bevacizumab) and Xeloda (Capecitabine) in Patients With Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18469
Record Dates: First submitted 2013-12-03; First posted 2013-12-17 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Bevacizumab; Capecitabine

ARMS (1):
- Avastin + Xeloda (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv on day 1 of each 3 week cycle.
Drug: capecitabine [Xeloda] — 1600mg/m2/day po in 2 divided doses, on days 1 to 14 of each 3 week cycle.

SUMMARY:
This study will evaluate the efficacy and safety of oral Xeloda (capecitabine) plus intravenous Avastin (bevacizumab) in patients with advanced or metastatic liver cancer. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* advanced or metastatic liver cancer;
* >=1 measurable lesion.

Exclusion Criteria:

* current radiotherapy, chemotherapy, or other experimental therapies;
* prior cytotoxic chemotherapy;
* major surgery, open biopsy, or traumatic injury within 28 days of study entry;
* history of a malignancy during the last 5 years, other than cutaneous basal cell cancer or in situ cervical cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Melbourne, Australia
- Hong Kong, Hong Kong
- Singapore, Singapore
- Taiwan (2):
  - Kueishan
  - Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab/Capecitabine: A cycle was defined as the following: Participants received 7.5 milligrams per kilogram (mg/kg) bevacizumab intravenously (IV) on Day 1; and 1600 mg per square meter per day (mg/m^2/day) capecitabine tablets, orally (PO), in a divided dose every 12 hours starting the evening of Day 1 and ending on the morning of Day 15, followed by 1 week of no treatment. This cycle was repeated every 3 weeks until disease progression, development of unacceptable toxicity, or for a maximum of 6 cycles. If all 6 cycles were tolerated without disease progression or development of unacceptable toxicity, participants then could have repeated the cycle until disease progression.
Period: Overall Study
Arm/Group | Bevacizumab/Capecitabine
Started | 45
Completed | 15
Not Completed | 30
Not completed — Adverse Event | 3
Not completed — Death | 1
Not completed — Insufficient therapeutic response | 25
Not completed — Refused treatment | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Bevacizumab/Capecitabine: A cycle was defined as the following: Participants received 7.5 mg/kg bevacizumab IV on Day 1 and 1600 mg/m^2/day capecitabine, tablets, PO, in a divided dose every 12 hours starting the evening of Day 1 and ending on the morning of Day 15, followed by 1 week of no treatment. This cycle was repeated every 3 weeks until disease progression, development of unacceptable toxicity, or for a maximum of 6 cycles. If all 6 cycles were tolerated without disease progression or development of unacceptable toxicity, participants then could have repeated the cycle until disease progression.
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. The best overall response achieved within the time from first drug administration to progressive disease or end of study was reported. CR was defined as complete disappearance of all target lesions and non-target disease, with the normalization of tumor marker levels. No new lesions. PR was defined as greater than or equal to (≥) 30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target lesions. Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker levels above the normal limits. No new lesions.
Time Frame: Screening; Weeks 6, 12, 18, 24, and 30; Every 3 months through follow-up
Population: Per Protocol (PP) Population included participants who: received greater than or equal to (≥) 1 dose of study medication, ≥6 weeks of treatment (unless excluded for allowed reasons), did not severely violate inclusion/exclusion criteria, had tumor assessment, greater than (>) 50% of first 6 weeks of treatment, and were not replaced.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 44
percentage of participants | 9.1 [2.5 to 21.7]

2. Secondary Outcome: Percentage of Participants With Disease Control
Description: The percentage of participants with disease control was based on assessment of confirmed CR, PR, or stable disease (SD) according to RECIST criteria. Confirmed responses were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. The best overall response achieved within the time from first drug administration to progressive disease or end of study was reported. CR was defined as complete disappearance of all target lesions and non-target disease, with the normalization of tumor marker levels. No new lesions. PR was defined as ≥ 30 % decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target lesions. Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker levels above the normal limits. No new lesions. SD was defined as not qualifying for PR or progressive disease.
Time Frame: Screening; Weeks 6, 12, 18, 24, and 30; Every 3 months through follow-up
Population: PP population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 44
percentage of participants | 52.3 [36.7 to 67.5]

3. Secondary Outcome: Time to Disease Progression - Percentage of Participants With an Event
Description: Time to progression was measured from time of treatment commencement to time of disease progression, or the date of death. Participants who were not progressed at the time of study completion (including participants who died before progressive disease) or who were lost to follow-up were censored at the date of last tumor assessment.
Time Frame: Screening; Weeks 6, 12, 18, 24, and 30; Every 3 months through follow-up
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 44
percentage of participants | 77.8

4. Secondary Outcome: Time to Disease Progression
Description: Time to progression was measured from time of treatment commencement to time of disease progression, or the date of death. Participants who were not progressed at the time of study completion (including participants who died before progressive disease) or who were lost to follow-up were censored at the date of their tumor assessment.
Time Frame: Screening; Weeks 6, 12, 18, 24, and 30; Every 3 months through follow-up
Population: Intent-To-Treat (ITT) Population included all enrolled participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 44
months | 2.8 [1.5 to 4.1]

5. Secondary Outcome: Time to Disease Progression - Percentage of Participants Progression-free at 12 Months
Description: as for outcome 3
Time Frame: Day 1, Weeks 1-18, Weeks 24 and 30, then every 3 months until death.
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 8
percentage of participants | 24.0 [11.0 to 37.0]

6. Secondary Outcome: Overall Survival - Percentage of Participants With an Event
Description: Overall Survival was defined as the time in months from randomization to date of death due to any cause. Participants without an event were censored the last time they were known to be alive.
Time Frame: Day 1, Weeks 1-18, Weeks 24 and 30, then every 3 months until death.
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 44
percentage of participants | 77.8

7. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time in months from randomization to date of death due to any cause. Participants without an event were censored the last time they were known to be alive. Median Overall Survival was estimated using the Kaplan-Meier method.
Time Frame: Day 1, Weeks 1-18, Weeks 24 and 30, then every 3 months until death.
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 44
months | 5.9 [4.1 to 9.7]

8. Secondary Outcome: Overall Survival - Percentage of Participants Event Free at 12 Months
Description: as for outcome 6
Time Frame: Day 1, Weeks 1-18, Weeks 24 and 30, then every 3 months until death.
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab/Capecitabine
Number analyzed (Participants) | 11
percentage of participants | 27 [14.0 to 40.0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from first intake of study medication until 28 days after the last intake of study medication with follow-up up until the event resolved or was adequately explained.
Description: Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.
Arm/Group | Bevacizumab/Capecitabine
Serious Adverse Events (participants affected / at risk) | 15/45
Other Adverse Events (participants affected / at risk) | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab/Capecitabine (N=45)
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Oedema peripheral (General disorders) | 1
Anal abscess (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hepatitis fulminant (Hepatobiliary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab/Capecitabine (N=45)
Diarrhoea (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal distention (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Bowel sounds abnormal (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 9
Fatigue (General disorders) | 6
Malaise (General disorders) | 5
Mucosal inflammation (General disorders) | 5
Chest discomfort (General disorders) | 3
Pain (General disorders) | 3
Chest pain (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Oedema (General disorders) | 1
Pitting oedema (General disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Weight decreased (Investigations) | 4
Haemoglobin (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Prostate examination abnormal (Investigations) | 1
Insomnia (Psychiatric disorders) | 7
Confusional state (Psychiatric disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Anal abscess (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Dysuria (Renal and urinary disorders) | 3
Haemorrhage urinary tract (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Jaundice (Hepatobiliary disorders) | 2
Hepatitis fulminant (Hepatobiliary disorders) | 1
Dry eye (Eye disorders) | 2
Keratitis (Eye disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Palpitations (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.